CLINICAL TRIAL: NCT00431587
Title: Changes in Different Fat Compartments During Weight Loss and Their Effect on Particular Manifestations of Metabolic Syndrome After Bariatric Procedures.
Brief Title: Changes in Different Fat Compartments and Their Effect on Particular Manifestations of Metabolic Syndrome After Bariatric Procedures.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hadassah Medical Organization (Other)
Other Study IDs: metabo-HMO-CTIL
Record Dates: First submitted 2007-02-05; First posted 2007-02-06 (Estimated); Last update posted 2008-04-17 (Estimated); Status verified 2007-01

CONDITIONS: Morbid Obesity; Metabolic Syndrome; Visceral Obesity
Keywords: morbid obesity; metabolic syndrome; visceral fat; peripheral fat
MeSH Terms: conditions — Obesity, Morbid; Metabolic Syndrome; Obesity, Abdominal

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The metabolic risks associated with obesity are closely correlated with central (abdominal), rather than a peripheral (gluteofemoral) fat pattern It has been shown that weight loss after bariatric surgery is followed by metabolic improvements.

The amount of fat lost from each site may be independently regulated. Very scant information is found in the literature regarding the relative changes in different fat body compartments, and their effect on the improvement of the metabolic profile.

In this study we define the absolute and relative changes in the different adipose tissue compartment after weight loss surgery

DETAILED DESCRIPTION:
The metabolic risks associated with obesity are closely correlated with central (abdominal), rather than a peripheral (gluteofemoral) fat pattern.

The amount of fat lost from each site may be independently regulated. Very scant information is found in the literature regarding the relative changes in different fat body compartments.

Rapid and preferential reduction of visceral fat mass could occur in morbid obese with visceral obesity. It has been previously shown, and it was also partially confirmed in this study, that a reduction in visceral fat was associated with metabolic improvements that included improved glucose tolerance and reduced plasma insulin and lipid levels.

This again suggests a threshold of proportional visceral fat loss, above which there is an improvement in insulin sensitivity and other component of metabolic syndrom.

We will quantify the different fat compartments changes after bariatric surgery by means of CT scan.

ELIGIBILITY:
Inclusion Criteria:

* Morbid obesity,
* Metabolic syndrome

Exclusion Criteria:

* Previous abdominoplasty surgery,
* Previous major abdominal surgey

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2007-06

CONTACTS AND LOCATIONS:
Overall Officials: Andrei Keidar, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization,, Jerusalem, Israel

REFERENCES:
- [Derived] Weiss R, Appelbaum L, Schweiger C, Matot I, Constantini N, Idan A, Shussman N, Sosna J, Keidar A. Short-term dynamics and metabolic impact of abdominal fat depots after bariatric surgery. Diabetes Care. 2009 Oct;32(10):1910-5. doi: 10.2337/dc09-0943. Epub 2009 Jul 8. PMID 19587363